CLINICAL TRIAL: NCT03672253
Title: Study of CAR-T Cells Targeting BCMA for Previously CAR-T Treated Refractory/Relapsed Multiple Myeloma
Brief Title: CAR-T Re-treatment for Refractory/Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T re-treatment-MM
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma Progression
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Re-treatment group (Experimental): Patients will be treated with CAR-T cells targeting BCMA (Different epitope with the previous CAR-T cell treatment they had been used) with a escalation approach, 0.5x10^6- 2.0x10^6 CAR-T cells/kg.
  Interventions: Drug: CAR-T Re-treatment

INTERVENTIONS:
Drug: CAR-T Re-treatment — Patients will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) or use their mononuclear cells that preserved in the laboratory for the production of CAR-T cells. After a pre-treatment lymphodepletion therapy, patients will receive the re-treatment of CAR-T therapy by intravenous injection.
  Other Names: CAR-T Re-treatment for r/r MM targeting BCMA

SUMMARY:
This is a single arm, open-label, single-center, phase 1 study, to determine the safety and efficacy of autologous reinfusion of CAR-T cells targeting BCMA in the treatment of refractory/relapsed multiple myeloma (r/r MM) who get recurrence and progression after previous CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed prior diagnosis of active multiple myeloma as defined by the updated IMWG criteria.
2. Patients with refractory multiple myeloma. Clear BCMA expression must be detected on malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry.
3. Refractory disease：1) At least 3 prior regimens, which must at least have contained bortezomi. or 2) other circumstances identified by clinical doctors.
4. Relapse criteria in NCCN clinical practice guidelines in Oncology: Multiple Myeloma (2016.V2).

Exclusion Criteria:

1. Women of child-bearing potential or who are pregnant or breastfeeding.
2. Have any active and uncontrolled infection: hepatitis B, hepatitis C, HIV, or other fatal viral and bacterial infection.
3. Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to either the required leukapheresis or the initiation of the conditioning chemotherapy regimen.
4. Patients with any uncontrolled intercurrent illness or serious uncontrolled medical disorder.
5. Patients with CNS metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions and spinal cord compression).
6. History of allogeneic stem cell transplantation. Have active acute or chronic graft-versus-host-disease (GVHD), or require immunosuppressant medications for GVHD, within 6 months of enrollment.
7. Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.
8. other conditions that excluded by clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events | Day 1-30 days after injection
  assessed by CTCAE v4.0, >= Grade 1 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-myeloma responses | Day 1-60 months
  by measuring the changes of aberrant immunoglobulin in serum
Anti-myeloma responses | Day 1-60 months
  multiple myeloma cells in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Hong Zhao, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided